CLINICAL TRIAL: NCT00387491
Title: A Randomized, Double-blind, 4-period Crossover, Dose-ranging Study to Determine the Effects on the Oral-cecal Transit Time of Single Doses of MOA-728 and the Safety and Tolerability of Multiple Doses of MOA-728 in Stable Methadone Maintenance Subjects
Brief Title: Dose Ranging Study in Healthy Methadone Maintenance Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Jeff Cohn, Salix Pharmaceuticals
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 3200A3-102
Record Dates: First submitted 2006-10-11; First posted 2006-10-13 (Estimated); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Adult

INTERVENTIONS:
Drug: MOA-728

SUMMARY:
To assess the effect of a single oral dose of MOA-728, an investigational drug, on the oral-cecal transit time in subjects who are taking methadone.

ELIGIBILITY:
1. Men or nonlactating and nonpregnant women, aged 18 to 65 years
2. Healthy as determined by the investigator on the basis of medical history, physical examination, clinical laboratory test results, vital signs, and 12-lead electrocardiogram

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16
Dates: Start 2006-06; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Oral-cecal transit time will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Cohn, Study Director — Bausch Health Americas, Inc.
Locations (1):
- Lenexa, Kansas, United States